CLINICAL TRIAL: NCT05482399
Title: Utility of Coronary Artery Calcification With Statin Therapy in Multimorbid Older Adults - An Ancillary Study Nested Within a Randomized Trial
Brief Title: STREAM Trial - Subclinical Atherosclerosis
Acronym: STREAM-SubATS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STREAM-SubATS; 32003B_205067 (Other Grant/Funding Number: Swiss National Science Foundation (SNSF)); FF21106 (Other Grant/Funding Number: Swiss Heart Foundation)
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Statin Treatment for Primary Prevention
Keywords: Coronary artery calcification; Statins; Primary prevention; Multimorbidity; Older adults

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study is open-label, with blinded outcome adjudication. Identification of potential outcome events is performed by blinded study team members. Participants, care providers, investigators and outcomes assessors are blinded to the baseline CAC scores.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Statin discontinuation (Experimental): Discontinuation of statin therapy - statin therapy will be stopped from the next scheduled intake after study inclusion (intervention arm).
  Interventions: Other: Statin discontinuation
- Statin continuation (No Intervention): Continuation of statin therapy - no change in the prescribed statin therapy (control arm).

INTERVENTIONS:
Other: Statin discontinuation — Statin therapy will be stopped. Additional lipid-lowering medication lowering LDL cholesterol will also be stopped.
  Other Names: Intervention arm
  Arms: Statin discontinuation

SUMMARY:
Statins are among the most widely used drugs. While they were found to be effective for primary and secondary prevention of cardiovascular disease (CVD) in middle-aged subjects, their benefits for primary prevention in older adults (aged ≥70 years) without CVD are uncertain, particularly for those with multimorbidity. To better target adults who may benefit from statins in primary prevention, coronary artery calcium (CAC) measurement is rapidly increasing in clinical use and is recommended for risk re-classification in some guidelines. Older patients with a high burden of subclinical atherosclerosis might benefit from continuing statins to prevent CV outcomes, but this hypothesis has not been rigorously tested in randomized clinical trials (RCTs). To address these questions, the investigators conduct a RCT in 500 multimorbid adults ≥70 years old taking statins for primary prevention who will be randomized to statin continuation vs. statin discontinuation, and measure baseline CAC to determine if the risk of a composite outcome of CV events and all-cause mortality after statin discontinuation differs among those with evidence of subclinical atherosclerosis at baseline as measured by CAC.

DETAILED DESCRIPTION:
Background & rationale: The benefit of statin use for primary prevention is uncertain in older adults with multimorbidity, while harms such as side effects may be more common in this population. Therefore, the 2018 AHA/ACC cholesterol guidelines mention that it may be reasonable to discontinue statins in multimorbid older adults without cardiovascular disease (CVD). To better target adults who may benefit from statins in primary prevention, coronary artery calcium (CAC) measurement is rapidly increasing in clinical use and is recommended for risk re-classification in some guidelines. Older patients with a high burden of subclinical atherosclerosis associated with cardiovascular (CV) risk might benefit from continuing statins to prevent CV outcomes, but this hypothesis has not been rigorously tested in randomized clinical trials (RCTs). To address this question, the investigators conduct a RCT in 500 multimorbid adults ≥70 years old taking statins for primary prevention who will be randomized to statin continuation vs. statin discontinuation, and measure baseline CAC to determine if the risk of a composite outcome of CV events and all-cause mortality after statin discontinuation differs among those with evidence of subclinical atherosclerosis at baseline as measured by CAC.

Specific aim:

To determine if the risk of a composite outcome of CV events and all-cause mortality after statin discontinuation differs among those with evidence of subclinical atherosclerosis at baseline as measured by CAC.

Design:

The study is a multicenter, randomized, non-inferiority trial conducted in multiple centers in Switzerland. Study subjects are randomly assigned in a 1:1 ratio to either discontinue (intervention arm) or continue (control arm) statin therapy. The study is open-label, with blinded outcome adjudication. After inclusion the study participants will be followed with phone calls, first after 3 months and then yearly for a mean of 24 months (min. follow-up period 12 months, max. follow-up period 48 months). Outcomes are assessed at each study follow-up. The investigators will use baseline native cardiac computed tomography scan to measure CAC to identify participants with subclinical atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* ≥70 years of age
* Multimorbid with ≥2 coexistent chronic conditions (defined by ICD-10 codes) with an estimated duration of 6 months or more based on clinical decision, besides dyslipidemia treated by statins
* Taking a statin for ≥80% of the time during the year before baseline

Exclusion criteria:

1. Secondary prevention based on previous large statin trials, defined as:

   * History of myocardial infarction type 12 (NSTEMI/STEMI) OR
   * History of unstable angina, defined as ACS symptomatic at rest, crescendo or new-onset angina (CCS 2 or 3) without ECG or cardiac biomarker changes (based on available documents) OR
   * Stable angina pectoris with a documented ischemia on a stress test or with a significant coronary disease defined as a coronary stenosis >50% OR
   * History of percutaneous coronary intervention (balloon or stent) or coronary artery bypass graft OR
   * History of ischemic stroke OR
   * History of Transient Ischemic Attack, defined as transient neurological deficit without diffusion restriction in MRI OR
   * History of carotid revascularization (stent or bypass) OR
   * History of peripheral arterial disease requiring revascularization (stent or bypass; Fontaine IV)
2. Aortic disease that required a vascular repair or aortic aneurysm with a maximum diameter >5.5 cm (men) or >5.2 cm (women) based on available documents
3. Diagnosis of familial hypercholesterolemia based on Dutch lipid score ≥6 based on available documents (LDL-c, Family History, Personal History)
4. Elevated risk of death within 3 months after baseline, defined as:

   * Hospitalized patients planned for palliative care within 24h of admission OR
   * Hospitalized patients with a Palliative Performance Scale (PPS) level <30% (based on situation at least 1 month before hospitalization), this corresponds to an estimated survival of 43% after 3 months; OR
   * Patients with an advanced metastatic cancer prognosis of ≤20% survival rate within 1 year after baseline (based on an online tool: https://cancersurvivalrates.com)
5. Body measures exceeding the CT scanner limits (morbid obesity exceeding weight and diameter limits)
6. Cardiac implants with metallic interference, such as pacemaker and mechanical heart valves
7. Orthopedic hardware in the mid or lower thoracic spine
8. Inability to hold breath for 10 seconds

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-06-21 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of all-cause death and major non-fatal CV events (non-fatal myocardial infarction, non-fatal ischemic stroke) | Up to 48 months
  The primary endpoint is a composite endpoint of all-cause death and major non-fatal CV events (non-fatal myocardial infarction, non-fatal ischemic stroke). All-cause death (and not CV death only) is chosen to account for a possible shift from CV to other causes of death. The composite endpoint was selected to assess the net clinical benefit in this population with expected high mortality. The clinical event committee which classifies suspected events for the primary and secondary clinical outcomes is blinded.

SECONDARY OUTCOMES:
All-cause death | Up to 48 months
  All deaths (for any reason)
Non-CV death | Up to 48 months
  All deaths except of deaths due to major CV events
Major CV events | Up to 48 months
  CV death, non-fatal myocardial infarction and non-fatal ischemic stroke
Total CV events | Up to 48 months
  CV death, non-fatal myocardial infarction, hospitalization for unstable angina, non-fatal ischemic stroke (including TIA) and arterial revascularization (coronary and peripheral urgent and non-urgent revascularization)
Total composite events | Up to 48 months
  All-cause death, non-fatal myocardial infarction, hospitalization for unstable angina, non-fatal ischemic stroke (including TIA) and arterial revascularization (coronary and peripheral urgent and non-urgent revascularization)
EQ-5D questionnaire | 3, 12 (primary analysis), 24, 36, 48 months
  EQ-5D is the name of the instrument and not an acronym. General quality of life assessment. The possible range of scores goes from 0 to 1.0, with higher scores indicating better quality of life.
Verbal numeric pain rating score (VNPRS) | 3 months
  To assess statin associated muscle symptoms. The VNPRS is an 11-point scale scored from 0-10, with higher scores indicating higher degree of pain.
Self-reported falls | Up to 12 months
  Self-reported falls, each participant will collect and list all falls during the first 12 months after randomization. Circumstances and medical consequences of each fall will be collected. Aggregated as rate of falls (falls per person per year).
Strength, assistance with walking, rising from a chair, climbing stairs, and falls (SARC-F questionnaire) | 12 (primary analysis), 24, 36, 48 months
  5-item questionnaire, the score ranges from 0 to 10 with higher scores indicating higher degree of sarcopenia.
Girerd medication adherence scale | 12 (primary analysis), 24, 36, 48 months
  6-item questionnaire, the score ranges from 0 to 6, higher scores indicating worse medication adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel R Blum, MD, MSc, Principal Investigator — University Hospital of Bern, University of Bern, Switzerland; Institute of Primary Health Care, University of Bern, Switzerland
Locations (1):
- University Hospital of Bern, University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Data will be deposited in the BORIS Research Data, the research data repository of the University of Bern. BORIS Research Data allows searching and is indexed by search engines. All items are stored with a unique Digital Object Identifier (DOI) that can be referenced in respective publication. It should be noted that the investigators plan to register and deposit data that relates to individual, primary publications and not the whole study database as such, as the investigators will use them for secondary analysis. This enables other researchers to replicate published analyses and results as well as to re-use the data for additional analyses such as metaanalysis.
  It is planned to disseminate the results of the trial to key target groups using the Lavis' framework for research knowledge transfer
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Foreseen for one year after publication of the main trial results. Items will be retained indefinitely.
Access Criteria: All efforts will be made to protect privacy and to de-identify the data. However, datasets contain sensitive data. Therefore, data will be shared on request under the following conditions:
  * A meaningful study question by the requester
  * Outline of the planned analyses
  * Valid methodology Signed data sharing agreement that contains a confidentiality agreement and other obligations to ensure privacy of trial participants
URL: https://boris.unibe.ch/policies.html